CLINICAL TRIAL: NCT06371703
Title: Enhancing Radiation Safety for Nuclear Medicine Radiographers: the Impact of Introducing the Automated Radiopharmaceutical Preparation and Administration System
Brief Title: Enhancing Radiation Safety for Nuclear Medicine Radiographers: the Impact of Introducing the Automat-ed Radiopharmaceutical Preparation and Administration System
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, PI, IRCCS San Raffaele
Other Study IDs: PETCT_INTEGO
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-04

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: automated system in reducing radiation exposure — evaluate the effectiveness of the automated system in reducing radiation exposure for radiographers involved in PET/CT procedures.

SUMMARY:
This project aims to evaluate the impact of the introduction of an automated system for radiopharmaceutical preparation and administration on the radiation safety of the radiographers working in nuclear medicine. This study will help to fill the existing gap in the scientific literature and provide useful guidance for the selection of the safest and most effective automated infusion system.

ELIGIBILITY:
Inclusion Criteria:

* 1)Nuclear medicine radiographers with experience in manual prepa-ration of radiopharmaceuticals.

  2) Nuclear medicine healthcare professionals with experience in radiopharmaceutical administration.

  3) Ability to provide written informed consent.

Exclusion Criteria:

* 1) Nuclear medicine radiographers without experience in manual preparation of radiopharmaceuticals.

  2) Nuclear medicine healthcare professionals without experience in radiopharmaceutical administration.

  3) Inability to provide written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals working in nuclear medicine departments
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in absorbed dose by radiographers during PET/CT procedures, measured in millisieverts (mSv). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Chiti, Study Director — IRCCS Ospedale San Raffaele
Locations (1):
- Irccs San Raffaele, Milan, Italy